CLINICAL TRIAL: NCT04210570
Title: Decreasing Environmental Impact and Costs of Using Inhalational Anesthetics by Replacing Chemical Absorbers With an Innovative Carbon Dioxide Membrane Filter System - a Prospective, Randomized, Clinical Trial
Brief Title: Decreasing Environmental Impact and Costs of Using Inhalational Anesthetic With a Carbon Dioxide Membrane Filter System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 114511
Record Dates: First submitted 2019-11-25; First posted 2019-12-24 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Anesthesia; Inhalation; Vapor
Keywords: Anesthesia; Inhalation; Vapour; CO2 Absorber; Minimal Flow Anesthesia; Memsorb; Healthcare Cost; Greenhouse gas; Environment Healthcare
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Memsorb GA (Experimental): Memsorb Filter will be used during general anesthesia (GA), fresh gas flow and ventilator settings are not modified
  Interventions: Device: Memsorb
- CGA GA (Active Comparator): Chemical CO2 absorber (CGA) will be used during general anesthesia (GA), fresh gas flow and ventilator settings are not modified
  Interventions: Drug: Chemical granulate absorber
- Memsorb low-flow (Experimental): Memsorb Filter will be used during low flow general anesthesia (GA)
  Interventions: Device: Memsorb
- CGA low flow (Experimental): Chemical CO2 absorber (CGA) will be used during low flow general anesthesia (GA)
  Interventions: Drug: Chemical granulate absorber
- Memsorb laparoscopic surgery (Experimental): Memsorb Filter will be used during general anesthesia for laparoscopic surgery
  Interventions: Device: Memsorb
- CGA laparoscopic surgery (Experimental): Chemical CO2 absorber (CGA) will be used during laparoscopic surgery
  Interventions: Drug: Chemical granulate absorber

INTERVENTIONS:
Device: Memsorb — Memsorb uses a polymeric membrane (similar to the ones used in oxygenators for cardiac surgery) that selectively allows CO2 to leave the rebreathing system while maintaining the inhalational anesthetic in the anesthesia circuit
  Arms: Memsorb GA; Memsorb laparoscopic surgery; Memsorb low-flow
Drug: Chemical granulate absorber — Chemical granulate absorber trap CO2 chemically in granules that are later disposed of when absorption capacity is reached
  Arms: CGA GA; CGA laparoscopic surgery; CGA low flow

SUMMARY:
Efficient inhalational anesthetic delivery requires the use of low-flow air and oxygen to reduce drug waste and minimize workspace contamination and environmental pollution. Currently, excess anesthetic gas is scavenged and removed from the operating room via the hospital ventilation system, where it is released into the atmosphere. CO2 is removed from the anesthesia circuit by the use of CO2 removal systems to prevent re-breathing and potential hypercarbia.

Carbon dioxide is currently removed using chemical granulate absorbers (CGAs), which trap CO2 in the granules that are later disposed of when absorption capacity is reached. They require replacement approximately every other day when used in moderate to high volume surgical centres, placing a costly burden on the healthcare system and environment (landfill).

One of the more concerning downfalls of using CGAs is the potential for the inhalational anesthetics to react with the granules and potentially produce toxic byproducts known as compounds A-E that are nephrotoxic and neurotoxic and require excess amounts of anesthetic gas to dilute.

This excess use of anesthetics gases places a financial burden on the healthcare system and has a detrimental impact on the environment. The vast majority of the gases used are eventually released into the environment with little to no degradation where they accumulate in the troposphere and act as greenhouse gases.

DMF Medical has created Memsorb, a new CO2 filtration membrane. Memsorb can remove CO2 from the anesthesia circuit without the use of CGAs, thereby eliminating the potential for toxic byproducts and allowing for significantly lower air and oxygen flow to be used, resulting in less use of inhalational anesthetics. Memsorb uses a polymeric membrane (similar to the ones used in oxygenators for cardiac surgery) that selectively allows CO2 to leave the rebreathing system, while maintaining the inhalational anesthetic in the circuit.

The lifespan of Memsorb is at least 12 months, resulting in less particulate waste and a decreased cost to the healthcare system.

We wish to evaluate the ability and efficacy of Memsorb in removing CO2 from the anesthesia circuit while maintaining physiologic minute volume ventilation, as compared to the traditional CGAs in a variety of surgical procedures, patient populations, and anesthesia gas flows.

ELIGIBILITY:
Inclusion Criteria:

* ASA I - III
* Elective surgical procedure
* Laparoscopic surgery for study aim III

Exclusion Criteria:

* ASA > IV
* Emergency surgery
* Severe respiratory disease (eg Asthma)
* Raised intracranial pressure
* Regional anesthesia
* Absence of arterial line for study aim III
* Self-reported pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of Memsorb compared to CGA to eliminate CO2 | Duration of general anesthesia (up to 12 hours)
  etCO2 (mmHg) and tidal volumes (ml) will be measured with the two systems in GE / Dates Ohmeda anesthesia machines
Impact of Memsorb, using minimal flow anesthesia (≤ 0.50 L/min), on the amount of inhalational anesthetic (ml) used, compared to standard practice | Duration of general anesthesia (up to 12 hours)
  Usage of Desflurane in ml will be measured during minimal flow (≤ 0.5 L/min) anesthesia, compared to traditional higher gas flow (> 2 L/min).
Effectiveness of using Memsorb during ventilation for removal of CO2 in laparoscopic surgeries resulting in high CO2 exposure, compared to CGAs | Duration of general anesthesia (up to 12 hours)
  etCO2 (mmHg), paCO2 (mmHg) and tidal volumes (ml) needed remove CO2 during laparoscopic surgery, resulting in higher CO2 exposure.

SECONDARY OUTCOMES:
Amount of inhaled anesthetics used | Duration of general anesthesia (up to 12 hours)
  Usage on inhaled anesthetics in ml for the surgery.
Duration of anesthesia | Duration of general anesthesia (up to 12 hours)
  Durantion measured in minutes
Water build up in anesthesia circuit | Duration of general anesthesia (up to 12 hours)
  Likert scale to measure water build up (1- no water, 3 - large amount of water)
Freshgas flow during general anesthesia | Duration of general anesthesia (up to 12 hours)
  Measured in ml/min
Number of CGAs used during the study period | Duration of general anesthesia (up to 12 hours)
  absolute number of canisters used
Minute volume ventilation | Duration of general anesthesia (up to 12 hours)
  tidal volume (ml) x respiratory rate (/min)

CONTACTS AND LOCATIONS:
Locations (1):
- LHSC, London, Ontario, Canada